CLINICAL TRIAL: NCT02101008
Title: Disulfiram and Chelated Zinc for the Rx of Disseminated Mets Mel That Has Failed First Line Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI37833
Record Dates: First submitted 2014-03-10; First posted 2014-04-01 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Disulfiram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Disulfiram and chelated zinc (Other): There is only one arm. All patients are treated wtih disulfiram and chelated zinc.
  Interventions: Drug: disulfiram and chelated zinc

INTERVENTIONS:
Drug: disulfiram and chelated zinc

SUMMARY:
Primary Objectives Determine the response rate associated with treatment of refractory disseminated malignant melanoma with disulfiram and chelated zinc.

Secondary Objectives Determine the progression-free survival associated with treatment of refractory disseminated malignant melanoma with disulfiram and chelated zinc.

Determine the overall survival associated with treatment of refractory disseminated malignant melanoma with disulfiram and chelated zinc.

Determine the toxicity associated with treatment of refractory disseminated malignant melanoma with disulfiram and chelated zinc Determine the effect of disulfiram and chelated zinc on in vivo protein S-glutathionylation.

ELIGIBILITY:
Inclusion Criteria:

The subjects must fulfill all the following inclusion criteria to be eligible for participation in the study, unless otherwise specified:

1. Male and female patients with stage IV melanoma cancer with biopsy proven metastases demonstrated by imaging studies. Extent of disease should be documented by CT scanning of the chest, abdomen and pelvis, or PET/CT scanning. At least one site of disease should be measurable by RECIST criteria.
2. Age of 18 years or more
3. ECOG performance status of 0 - 2
4. Patients must have received and progressed after or not responded to at least one cycle of first line therapy (chemotherapy, biotherapy, or biochemotherapy) or are unwilling or ineligible to undergo standard therapy
5. Patients with brain metastases along with disease at other sites are eligible to participate if their brain disease has been treated with surgery or radiation
6. Not currently receiving other cancer chemotherapy
7. Not currently participating in another study
8. Baseline AST and ALT not greater than 2.0 X upper limit of normal
9. Able and willing to provide informed consent and to comply with study procedures
10. Able to ingest oral medications
11. No known allergy to disulfiram or zinc gluconate
12. Willing to refrain from ingestion of alcoholic beverages while on the study
13. Serum copper within the normal range at baseline, or if outside the normal range, the PI will review for clinical significance

Exclusion Criteria:

Potential study subjects who meet any of the following criteria are not eligible for participation in the study:

1. Participation in another clinical trial of a therapeutic drug during the past 30 days
2. Addiction to alcohol or cocaine
3. Baseline AST or ALT greater than 2.0 X upper limit of normal
4. Unable to ingest oral medications
5. Unable to undergo CT scanning because of inability to lie recumbent in the scanner;
6. Actively receiving cytotoxic cancer chemotherapy agents
7. Evidence of thiuram allergy (may present as contact allergy to rubber or elastic)
8. Current use of sertraline and cyclosporine
9. Women of child-bearing potential who are not using a commonly accepted effective means of contraception; women of child-bearing potential will have a pregnancy test before enrollment
10. Need for warfarin or theophylline, the metabolism of which is likely influenced by disulfiram
11. Pregnant women and nursing mothers are not allowed to enroll on this study
12. Patients who are taking medications metabolized by cytochrome P450 2E1, including chlorzoxazone or halothane and its derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2013-02 (Actual); Study Completion 2013-11-27 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Disulfiram and Chelated Zinc: There is only one arm. All patients are treated wtih disulfiram and chelated zinc. Disulfiram will be administered at a fixed dose of 250 mg orally per day at bedtime. Chelated zinc will be given at a dose of 50 mg orally 3 times a day (with each meal).
Period: Overall Study
Arm/Group | Disulfiram and Chelated Zinc
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Disulfiram and Chelated Zinc: There is only one arm. All patients are treated wtih disulfiram and chelated zinc.
  disulfiram and chelated zinc
Arm/Group | Disulfiram and Chelated Zinc
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 65 [52 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate to Treatment of Melanoma With Disulfiram and Chelated Zinc
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT scanning of the chest, abdomen and pelvis, or PET/CT scanning.: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Response to treatment will be measured by RECIST evaluation at disease assessment time-points from date of randomization until the date of first documented progression or death from any cause whichever came first (up to 15 months.)
Measure: Number; unit: participants
Arm/Group | Disulfiram and Chelated Zinc
Number analyzed (Participants) | 12
participants | 0

2. Secondary Outcome: Progression Free Survival
Time Frame: Every 56 days - for up to two years
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Disulfiram and Chelated Zinc
Number analyzed (Participants) | 12
days | 51.8 (39.8)

ADVERSE EVENTS:
Arm/Group | Disulfiram and Chelated Zinc
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Disulfiram and Chelated Zinc (N=12)
Confusion (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Disulfiram and Chelated Zinc (N=12)
Fatigue (General disorders) | 7
rash (Infections and infestations) | 2
pruritis (Skin and subcutaneous tissue disorders) | 2
diarrhea (Gastrointestinal disorders) | 3
nausea (Gastrointestinal disorders) | 4
consitpation (Gastrointestinal disorders) | 1
vomiting (Gastrointestinal disorders) | 1
dysgeusia (Nervous system disorders) | 2
Aspartate aminotransferase (Investigations) | 1
Alanine aminotransferase (Investigations) | 1
ataxia (Nervous system disorders) | 2
tremor (Nervous system disorders) | 1
confusion (Psychiatric disorders) | 4
headache (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
renal insufficiency (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes